CLINICAL TRIAL: NCT04987983
Title: A Comparison Study of the Bottle-feeding of Prematurely Born Infants (≤ 34 Weeks of Gestational Age) in Side-lying Position, Positioned on the Right and Left Side - a Pilot Study.
Brief Title: A Comparison Study of Feeding Prematures in the Side-lying Position on the Right and Left Side - a Pilot Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Polish Mother Memorial Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Anna Raczyńska, Principal Investigator, Polish Mother Memorial Hospital Research Institute
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: PMMHRI-2021
Record Dates: First submitted 2021-07-14; First posted 2021-08-03 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Bottle Feeding; Premature
Keywords: Premature Infant; Bottle Feeding; Side-lying Position; Oral Feeding
MeSH Terms: conditions — Bottle Feeding; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental SLP-R (Experimental): Infant placed in a SLP-R on the researcher's lap. Infant body positioned on side-lying position on the right side of it's body. Head of the infant symmetrically placed between the shoulders, supported by the researcher's. Shoulder girdle higher than the pelvic girdle, head and back in a straight line - a slight natural bend of the body is allowed. Legs bent at an angle of approx. 90° in the natural flexion of the knee and ankle joint. The infant's arms close to the midline (on the bottle or researcher's hands)
  Interventions: Other: Experimental SLP-R
- Experimental SLP-L (Experimental): Infant placed in a SLP-L on the researcher's lap. Infant body positioned on side-lying position on the left side of it's body. Head of the infant symmetrically placed between the shoulders, supported by the researcher's. Shoulder girdle higher than the pelvic girdle, head and back in a straight line - a slight natural bend of the body is allowed. Legs bent at an angle of approx. 90° in the natural flexion of the knee and ankle joint. The infant's arms close to the midline (on the bottle or researcher's hands).
  Interventions: Other: Experimental SLP-L

INTERVENTIONS:
Other: Experimental SLP-R — SLP-R will be given to the infant during bottle-feeding.
  Arms: Experimental SLP-R
Other: Experimental SLP-L — SLP-L will be given to the infant during bottle-feeding.
  Arms: Experimental SLP-L

SUMMARY:
Methods and techniques to improve the quality and safety of oral feeding in preterm infants are still a significant challenge in modern neonatology. One of the areas that can help improve feeding is choosing the optimal feeding position for premature babies.

DETAILED DESCRIPTION:
PURPOSE: The aim of the study is to compare the advantages of side-lying positioning on the right (SLP-R) and left side (SLP-L) of infant's body, during bottle-feeding of preterm infants.

METHOD: The study will include eight neonates (n=8) born ≤34 weeks of gestational age. Four bottle-feeding sessions will be tested in each of the newborns: two in the SLP-R and two in the SLP-L. The position for the first study will be randomly assign, then positioning will be change after each feeding session. In one day, only two consecutive feeding sessions will be tested which will be included to the study in order to minimize fatigability as a disrupting factor. The levels of saturation (SpO2) and heart rate (HR) will be measured as the parameters indicative of the newborn's physiological stability. The factors determining the qualitative aspect of feeding include the total time of declines of SpO2 ≤85%, level of the newborn's alertness according to the Neonatal Behavioral Assessment Scale (NBAS), and the occurrence of choking episodes. The proportion of milk consumed (volume of milk eaten relative to the expected volume) and the duration of the feeding and feeding session were also will be record. Maximum time of feeding session will be 40 minutes.

Also the posseting during/after feeding and regurgitations will be record in each tested positions.

ELIGIBILITY:
Inclusion Criteria:

* circulatory and respiratory stability;
* readiness for oral feeding according to each child's Speech-Language Pathologist assessment;
* prematurely born infants who will be in the process of transfer from enteral nutrition to full oral feeding and will be fed orally at least 4 times within twenty-four hours;
* researcher must be a right handed person (right hand is the dominant hand);
* each infant will be fed with one kind of bottle and nipple;
* parents will give a informed consent to participate their infant in the study.

Exclusion Criteria:

* disorders which could significantly affect the feeding course, such as cleft lip and/or palate, facial paralysis and/or congenital defects of the facial skeleton;
* the presence of detected congenital abnormalities and metabolic diseases;
* newborns after abdomen chirurgical treatment;
* low Apgar score (less than 5 points at the 5th and 10th minute of the measurement);
* administered analgesics, anticonvulsants and sedatives <72 hours from extubation prior the trial;
* parenterally fed infants;
* infants with administered intravenous infusion with glucose;
* parents refusal to participate in the study or when bottle-feeding will not be the parental preference.

Ages: 32 Weeks to 38 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2021-09-23 (Actual)

PRIMARY OUTCOMES:
Physiological stability | Measured 2 minutes before feeding session, in 3rd and 10th minutes of feeding, at the moment of finish of the feeding and in 10th minute after feeding (5 points of measurement)
  Oxygen saturation (SpO2) changes measured by using a pulse oximeter data
Physiological stability | Measured 2 minutes before feeding session, in 3rd and 10th minutes of feeding, at the moment of finish of the feeding and in 10th minute after feeding (5 points of measurement)
  Heart rate (HR) changes measured by using a pulse oximeter data
Qualitative aspect of bottle-feeding | Up to 40 minutes - measured during feeding session (maximum time of feeding session is 40 minutes)
  Total time of declines of SpO2 ≤85% measured by using a pulse oximeter data
Qualitative aspect of bottle-feeding | Measured 2 minutes before feeding session, in 3rd and 10th minutes of feeding, at the moment of finish of the feeding and in 10th minute after feeding (5 points of measurement)
  Level of the newborn's alertness changes according to the 6-point Neonatal Behavioral Assessment Scale, where individual points mean: 1 - quiet sleep, 2 - active sleep, 3 - drowsy, 4 - quiet alert, 5 - active alert, 6 - crying. This is descriptive, qualitative scale which shows changes of newborn's activity.
Qualitative aspect of bottle-feeding | Up to 40 minutes - measured during feeding session (maximum time of feeding session is 40 minutes)
  Occurrence of choking episodes
Qualitative aspect of bottle-feeding | Up to 40 minutes - measured during feeding session (maximum time of feeding session is 40 minutes)
  Occurence of posseting and regurgitations
Qualitative aspect of bottle-feeding | Up to 1 hour - measured from taking the baby out of bed before feeding to putting the baby to bed immediately after the intervention. Putting baby on parent's chest to kangaroo (Kangaroo Mother Care) after feeding instead to bed was also allowed.
  Duration of the feeding session
Qualitative aspect of bottle-feeding | Up to 40 minutes - measured during feeding session (maximum time of feeding session is 40 minutes) - measured from insertion of the nipple to the infant's mouth to the moment when baby finish the feeding
  Duration of feeding
Qualitative aspect of bottle-feeding | Up to 40 minutes - measured during feeding session (maximum time of feeding session is 40 minutes) - duration of feeding is measured from insertion of the nipple to the infant's mouth to the moment when baby finish the feeding
  Duration of feeding
Qualitative aspect of bottle-feeding | Measured in 10th minute of feeding and on the finish of the feeding - maximum in 40th minute of feeding (maximum time of feeding is 40 minutes)
  Proportion of milk consumed (volume of milk eaten relative to the expected volume)

CONTACTS AND LOCATIONS:
Overall Officials: Anna D Raczyńska, PhD, Principal Investigator — Polish Mother's Memorial Hospital - Research Institute
Locations (1):
- Polish Mother's Memorial Hospital - Research Institute, Lodz, Poland

IPD SHARING:
Plan to Share IPD: No